CLINICAL TRIAL: NCT03707795
Title: Treatment of FUS-Related ALS With Betamethasone - The TRANSLATE Study
Acronym: TRANSLATE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Edward Kasaraskis (Other)
Responsible Party: Sponsor-Investigator, Edward Kasaraskis, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-0159-F6A
Record Dates: First submitted 2017-09-14; First posted 2018-10-16 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Familial Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — betamethasone sodium phosphate; betamethasone acetate

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants remain blinded as to their genotype.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 - Amyotrophic Lateral Sclerosis (Experimental): Betamethasone sodium phosphate/betamethasone acetate (Celestone® Soluspan®), 30 mg IM once a day for four days
  Interventions: Drug: Betamethasone sodium phosphate/betamethasone acetate (Celestone® Soluspan®), 30 mg IM once a day for four days
- Arm 2 - Familial Amyotrophic Lateral Sclerosis (Active Comparator): Betamethasone sodium phosphate/betamethasone acetate (Celestone® Soluspan®), 30 mg IM once a day for four days
  Interventions: Drug: Betamethasone sodium phosphate/betamethasone acetate (Celestone® Soluspan®), 30 mg IM once a day for four days

INTERVENTIONS:
Drug: Betamethasone sodium phosphate/betamethasone acetate (Celestone® Soluspan®), 30 mg IM once a day for four days — Participants will be given four IM injections throughout the study

SUMMARY:
By doing this study the investigator hopes to learn more about a potential cause of amyotrophic lateral sclerosis (ALS) called "oxidative stress". Oxidative stress is essentially an imbalance between the production of certain chemicals in the body called "free radicals" and the ability of the body to counteract or detoxify their harmful effects through neutralization by antioxidants. It is thought that factors such as environmental exposure (chemicals and lead), diet, smoking,alcohol consumption, physical activity and psychological stress cause oxidative stress to occur inside the body.

By doing this study, the investigator hopes to learn whether the FDA-approved steroid medication called Betamethasone will restore overall antioxidant activity fALS patients with mutations in the Fused in Sarcoma gene (FUS gene).

Participants who agree to take part in this research study, agree to the following responsibilities:

* Attend all scheduled visits
* Notify the study doctor of any illnesses, unexpected or troublesome side effects, or any other medical problems that occur during the study
* Be completely honest with their answers to all questions
* Check with the study doctor before taking any new medications, whether prescribed or "over the counter," even vitamins and herbal supplements.

DETAILED DESCRIPTION:
This will be a single-blinded, pharmacokinetic and pharmacodynamics study of intramuscular (IM) betamethasone in ALS patients and non-ALS relatives from families with a mutation in the FUS gene. Participants remain blinded as to their genotype.

Betamethasone is a FDA-approved drug and is only available in an IM dosing form (Celestone®). This will be a proof-of-concept translational study built on discoveries made by our research team at the University of Kentucky. All participants will receive active drug.

The research procedures will be conducted at the University of Kentucky (UK) Albert B. Chandler Hospital, Pavilion H, 800 Rose Street, Lexington, KY. Participants will need to come to Center for Clinical and Translational Science (CCTS) on the 3rd Floor (Room C300) of Pavilion H, at UK Albert B. Chandler Hospital, for a Consent/Screening Visit. If found eligible and qualify for the study, participants will be asked to give voluntary written consent to participate.

Following signing the consent form, participants will be admitted to the UK Albert B. Chandler Hospital, CCTS Inpatient Unit, 5th Floor, 5 North Wing of the Hospital for 2 nights (approximately 48 hours). The following tests and procedures will take place:

* Neurological Exam
* Vital Signs (blood pressure, heart rate and respiratory rate) will be measured
* Medical and medication history will be collected
* Questionnaire
* blood specimen for Pharmacokinetic and Pharmacodynamic will be collected testing*
* Participants will also be asked to do some testing of their breathing and physical abilities.

The study drug (betamethasone sodium phosphate/betamethasone acetate [Celestone® Soluspan®]) will be injected into a muscle such as arm or buttock - this will be the first of the four injections of the study drug administered during the study.

At 24 hours after the first injection with the study drug, and while still in the the hospital, the study drug will again be injected into a muscle such as arm or buttock - this will be the second of the four injections of the study drug administered during the study.

Following this second treatment, and after the study doctor determines it is safe, the participant will be discharged from the hospital. They will will stay in a local motel overnight, awaiting the next day's blood draw, assessments, testing and 3rd treatment with study drug.

Participants who do not live close to the hospital, motel accommodations will be provided at no charge, for an overnight stay between the 48 Hour visit, and the 72 Hour scheduled follow-up visit.

At 72 hours after first injection with the study drug, the study drug will again be injected into a muscle such as arm or buttock - this will be the fourth and last of the four injections administered during the study. Following this fourth treatment, and after the study doctor determines if is safe, participants will be allowed to leave.

The 72 Hour (Day 3), 168 Hour (Day 7) and 336 Hour (Day 14) visits will take about 1 hour each. The approximate, total amount of time participants will be asked to volunteer for this study is 51 hours over the 336 hour (14 day) duration of this research study.

Participants or their insurance company, Medicare or Medicaid will be responsible for the costs of all routine medical care and treatment they would normally receive for their condition. The University of Kentucky may not be allowed to bill insurance companies, Medicare or Medicaid for the medical procedures done strictly for research.

Neither the participant or their provider will be charged for costs of any of the procedures performed for the research study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of familial ALS (fALS)
* Relative of a fALS person and carry the FUS gene

Exclusion Criteria:

* Under 20 years or over 80 years of age
* Cannot tolerate steroids, including betamethasone
* Are unwilling or unable to attend all scheduled research visits
* Currently participating in another clinical drug trial
* Major neurological disease, other than ALS
* Pregnant

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Betamethasone plasma levels | 14 days
  Blood will be collected at multiple time points (baseline, 24 hours, 48 hours, 72 hours, day 7 and day 14) for analysis of Betamethasone levels. Data will be reported as the change in Betamethasone over time.

SECONDARY OUTCOMES:
Protein carbonyl plasma levels | 14 days
  Blood will be collected at multiple time points (baseline, 24 hours, 48 hours, 72 hours, day 7 and day 14) for analysis of Protein carbonyl levels. Data will be reported as the change in Protein carbonyl over time.
Superoxide dismutase plasma levels | 14 days
  Blood will be collected at multiple time points (baseline, 24 hours, 48 hours, 72 hours, day 7 and day 14) for analysis of Superoxide dismutase levels. Data will be reported as the change in Superoxide dismutase over time.
Peroxide plasma levels | 14 days
  Blood will be collected at multiple time points (baseline, 24 hours, 48 hours, 72 hours, day 7 and day 14) for analysis of Peroxide levels. Data will be reported as the change in Peroxide over time.
Glutathione disulfide plasma levels | 14 days
  Blood will be collected at multiple time points (baseline, 24 hours, 48 hours, 72 hours, day 7 and day 14) for analysis of Glutathione disulfide levels. Data will be reported as the change in Glutathione disulfide over time.
Glutathione plasma levels | 14 days
  Blood will be collected at multiple time points (baseline, 24 hours, 48 hours, 72 hours, day 7 and day 14) for analysis of Glutathione disulfide levels. Data will be reported as the change in Glutathione disulfide over time.

OTHER OUTCOMES:
Slow vital capacity | 14 days
  Participants will blow into a spirometer at a natural rate of exhale to measure the vital capacity of their respratory system. Data will be reported as the change in vital capacity over time.
Maximum voluntary ventilation (MVV) | 14 days
  Participants will inhale as deeply and quickly as possible into a spirometerr to over the course of 15 seconds to assess respiratory function. Data will be reported as the change in MMV over time.
Grip strength | 14 days
  Participants will squeeze a dynamometer which will measure the maximal force generated in mmHG. Data will be reported as the change in grip strength over time.
Manual dexterity | 14 days
  Participants will have their gross movements of their arms, hands and fingers and their fine motor capacities measured using the Purdue Pegboard assessment. The test involves the placement of small pegs in a board at varying ranges of extremity extension. Participants are scored on the number of pegs they can place in a 30 second assessment. Data are presented as the change in number of pegs placed over time.
Sit to stand assessment | 14 days
  Participants will be timed in their ability to rise from a seated position to standing fully upright. Data are presented as the change in time to rise over time.
Time walk assessment | 14 days
  Participants will be time in their ability to walk 20 feet. Data are presented as the change in time to cover the distance over time.
Isometric strength generation | 14 days
  Utilizing an Accurate Test of Limb Isometric Strength (ATLIS) participants will their static isometric limb strength measured. Data are presented as the change in limb strength over time.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Kasarskis, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No